CLINICAL TRIAL: NCT05054257
Title: Safety and Efficacy of Anti-CD19 Chimeric Antigen Receptor-modified Autologous T Cells (CART19) in Patients with Relapsed/refractory CD19+ Acute Lymphoblastic Leukemia and Non-Hodgkin's Lymphoma. a Dose Escalation, Open-label, Phase I Study.
Brief Title: CART19 Cells Effects in Patients with Relapsed or Refractory Acute Lymphoblastic Leukemia and Non-Hodgkin's Lymphoma
Acronym: UHKT-CAR19-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology and Blood Transfusion, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHKT-CAR19-01; 2018-004789-32 (EudraCT Number)
Record Dates: First submitted 2021-07-19; First posted 2021-09-23 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma Refractory; Non-Hodgkin's Lymphoma, Relapsed
Keywords: B Cell; ALL; Relapsed or Refractory; B-NHL; Leukemia; Chimeric antigen receptor; CAR; CAR T cell
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CAR19 T lymphocytes (Experimental): Human Autologous T Lymphocytes Expressing the Chimeric Antigen Receptor Specific to CD19
  Interventions: Drug: Autologous CAR19 T lymphocytes

INTERVENTIONS:
Drug: Autologous CAR19 T lymphocytes — First-in-human trial examining the safety and efficacy of CART19 in r/r B-ALL and B-NHL

SUMMARY:
Phase I Dose Escalation Study of CART19 Cells for Adult Patients With Relapsed / Refractory Acute Lymphoblastic Leukemia and Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This is an open-label, single arm study on up to 24 adult subjects with refractory or relapsed CD19+ Non-Hodgkin's Lymphoma or B-ALL. Following lymphodepleting conditioning regimen, the patients will receive a single dose of autologous CAR19 T lymphocytes provided by the sponsor´s manufacturing facility. CART19 dose will be escalated in consecutive patients using accelerated titration design in order to establish recommended CART19 dose for further study, which will be either Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD), whichever is reached first.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with refractory or relapsing CD19 positive B-ALL or B-NHL defined as:

   1. B-ALL refractory to treatment or in the second or subsequent relapse (hematological OR molecular), OR
   2. B-NHL refractory to treatment or in first relapse ineligible for autologous stem cell transplantation (ASCT) or in second to fourth relapse, OR
   3. B-ALL or B-NHL relapsing after autologous or allogeneic hematopoietic cell transplantation (HCT).
2. CD19 expression on malignant cells confirmed by flow cytometry or by immunohistochemistry.
3. Age ≥18 years and ≤ 80 yearss.
4. Patient able to understand and sign informed consent.
5. Women of child-bearing potential: negative pregnancy test at enrolment (PSV) and at Visit 1.

General Exclusion Criteria:

1. Known hypersensitivity to any component of the Investigational Medicinal Product (IMP).
2. Autologous or allogeneic HCT in 3 months prior to IMP administration.
3. Severe, uncontrolled active infection.
4. Life expectancy < 6 weeks.
5. Parenchymal central nervous system involvement.
6. Respiratory insufficiency (need for oxygen therapy).
7. Significant liver impairment: bilirubin > 50 µmol/L, AST or ALT > 4times normal upper limit.
8. Acute kidney injury with serum creatinine > 180 µmol/L, oliguria or need for acute dialysis.
9. Heart failure with EF < 30% by echocardiography.
10. Presence of active grade 3-4 acute GvHD.
11. Serious uncontrolled neurological comorbidity.
12. Vaccination with live virus vaccines in the 4 weeks before IMP administration and within 90 days after the IMP dose.
13. Women: pregnancy or breast-feeding.
14. Subjects of fertile age, unless permanent sexual abstinence is their lifestyle choice:

    * female patients of childbearing potential not willing to use a highly effective method of contraception during the study,
    * male patients whose sexual partner(s) are women of childbearing potential who are not willing to use a highly effective method of contraception during the study.

Exclusion criteria to Procurement of IMP manufacture starting material

1. Severe uncontrolled active infection.
2. Positive test results for HIV1/2, Hepatitis B/C and lues.
3. Concurrent or recent prior therapies before apheresis:

   * Autologous or allogeneic hematopoietic cell transplantation within 12 weeks.
   * Clofarabine, Fludarabine, Alemtuzumab within 8 weeks.
   * Donor lymphocyte infusions within 4 weeks.
   * Pegylated asparaginase within 4 weeks.
   * Maintenance chemotherapy within 2 weeks.
   * Long-acting Granulocyte Colony Stimulating Factor (G-CSF) within 2 weeks.
   * Vincristine within 2 weeks.
   * Intrathecal methotrexate within 1 week.
   * Granulocyte Colony Stimulating Factor (G-CSF) within 5 days.
   * Therapeutic dose of corticosteroids within 3 days.
   * Short-acting cytostatics within 3 days

Exclusion criteria to IMP administration

1. Severe, uncontrolled active infections.
2. Life expectancy < 6 weeks.
3. Parenchymal central nervous system involvement
4. Respiratory insufficiency (need for oxygen therapy).
5. Significant liver impairment: bilirubin > 50 µmol/L, Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 4times normal upper limit.
6. Acute kidney injury with serum creatinine > 180 µg/L, oliguria or need for acute dialysis.
7. Heart failure with Ejection Fraction (EF) < 30% by echocardiography.
8. Presence of active grade 3 - 4 acute GvHD
9. Serious uncontrolled neurological comorbidity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years post treatment
  Cumulative incidence of IMP-related adverse events (AEs) graded by ASTCT consensus grading criteria for Cytokine Release Syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) and by Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 for other AEs. Toxicities will be followed from the start of Blood Collection or Apheresis until the end of the study.
Assessment of Dose-Limiting Toxicities (DLTs) | Up to 28 days after IMP administration
  Incidence of Dose-limiting toxicities (DLTs) during the first 28 days after IMP administration

SECONDARY OUTCOMES:
Complete remission ( CR) rate | CR rate at 100 days and 6 months after IMP administration
  Assessment of the efficacy of IMP cells administration in patients with refractory or relapsed CD19+ NHL and B-ALL evaluated by Complete Remission rate
Overall Survival | OS at 1 year after IMP administration
  Assessment of the efficacy of IMP cells administration in patients with refractory or relapsed CD19+ NHL and B-ALL evaluated by Overall Survival
Quality of life using the European Organization for the Research and Treatment of Cancer 30 item questionnaire (EORTC QLQ-C30). | At 6 months and 1 year following IMP administration
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small. A change of 10 - 20 points is considered a moderate change.

OTHER OUTCOMES:
CART19 cells in peripheral blood, bone marrow and cerebrospinal fluid | Up to 24 months
  Assessment of quantity and phenotype of CART19 cells in peripheral blood, bone marrow and cerebrospinal fluid using using flow-cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Petr Lesny, Study Chair — Institute of Hematology and Blood Transfusion, Czech Republic; Jan Vydra, Principal Investigator — Institute of Hematology and Blood Transfusion, Czech Republic
Locations (1):
- Institute of Hematology and Blood Transfusion, Czech Republic, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maude SL, Frey N, Shaw PA, Aplenc R, Barrett DM, Bunin NJ, Chew A, Gonzalez VE, Zheng Z, Lacey SF, Mahnke YD, Melenhorst JJ, Rheingold SR, Shen A, Teachey DT, Levine BL, June CH, Porter DL, Grupp SA. Chimeric antigen receptor T cells for sustained remissions in leukemia. N Engl J Med. 2014 Oct 16;371(16):1507-17. doi: 10.1056/NEJMoa1407222. PMID 25317870
- [Background] Porter DL, Hwang WT, Frey NV, Lacey SF, Shaw PA, Loren AW, Bagg A, Marcucci KT, Shen A, Gonzalez V, Ambrose D, Grupp SA, Chew A, Zheng Z, Milone MC, Levine BL, Melenhorst JJ, June CH. Chimeric antigen receptor T cells persist and induce sustained remissions in relapsed refractory chronic lymphocytic leukemia. Sci Transl Med. 2015 Sep 2;7(303):303ra139. doi: 10.1126/scitranslmed.aac5415. PMID 26333935
- [Background] Hartmann J, Schussler-Lenz M, Bondanza A, Buchholz CJ. Clinical development of CAR T cells-challenges and opportunities in translating innovative treatment concepts. EMBO Mol Med. 2017 Sep;9(9):1183-1197. doi: 10.15252/emmm.201607485. PMID 28765140
- [Background] Hamada M, Nishio N, Okuno Y, Suzuki S, Kawashima N, Muramatsu H, Tsubota S, Wilson MH, Morita D, Kataoka S, Ichikawa D, Murakami N, Taniguchi R, Suzuki K, Kojima D, Sekiya Y, Nishikawa E, Narita A, Hama A, Kojima S, Nakazawa Y, Takahashi Y. Integration Mapping of piggyBac-Mediated CD19 Chimeric Antigen Receptor T Cells Analyzed by Novel Tagmentation-Assisted PCR. EBioMedicine. 2018 Aug;34:18-26. doi: 10.1016/j.ebiom.2018.07.008. Epub 2018 Aug 3. PMID 30082227
- [Background] Tipanee J, VandenDriessche T, Chuah MK. Transposons: Moving Forward from Preclinical Studies to Clinical Trials. Hum Gene Ther. 2017 Nov;28(11):1087-1104. doi: 10.1089/hum.2017.128. Epub 2017 Aug 22. PMID 28920716
- [Background] Kebriaei P, Singh H, Huls MH, Figliola MJ, Bassett R, Olivares S, Jena B, Dawson MJ, Kumaresan PR, Su S, Maiti S, Dai J, Moriarity B, Forget MA, Senyukov V, Orozco A, Liu T, McCarty J, Jackson RN, Moyes JS, Rondon G, Qazilbash M, Ciurea S, Alousi A, Nieto Y, Rezvani K, Marin D, Popat U, Hosing C, Shpall EJ, Kantarjian H, Keating M, Wierda W, Do KA, Largaespada DA, Lee DA, Hackett PB, Champlin RE, Cooper LJ. Phase I trials using Sleeping Beauty to generate CD19-specific CAR T cells. J Clin Invest. 2016 Sep 1;126(9):3363-76. doi: 10.1172/JCI86721. Epub 2016 Aug 2. PMID 27482888
- [Background] Otahal P, Prukova D, Kral V, Fabry M, Vockova P, Lateckova L, Trneny M, Klener P. Lenalidomide enhances antitumor functions of chimeric antigen receptor modified T cells. Oncoimmunology. 2015 Dec 3;5(4):e1115940. doi: 10.1080/2162402X.2015.1115940. eCollection 2016 Apr. PMID 27141398
- [Background] Yusa K, Zhou L, Li MA, Bradley A, Craig NL. A hyperactive piggyBac transposase for mammalian applications. Proc Natl Acad Sci U S A. 2011 Jan 25;108(4):1531-6. doi: 10.1073/pnas.1008322108. Epub 2011 Jan 4. PMID 21205896
- [Background] Ptackova P, Musil J, Stach M, Lesny P, Nemeckova S, Kral V, Fabry M, Otahal P. A new approach to CAR T-cell gene engineering and cultivation using piggyBac transposon in the presence of IL-4, IL-7 and IL-21. Cytotherapy. 2018 Apr;20(4):507-520. doi: 10.1016/j.jcyt.2017.10.001. Epub 2018 Feb 21. PMID 29475789
- [Background] Milone MC, Fish JD, Carpenito C, Carroll RG, Binder GK, Teachey D, Samanta M, Lakhal M, Gloss B, Danet-Desnoyers G, Campana D, Riley JL, Grupp SA, June CH. Chimeric receptors containing CD137 signal transduction domains mediate enhanced survival of T cells and increased antileukemic efficacy in vivo. Mol Ther. 2009 Aug;17(8):1453-64. doi: 10.1038/mt.2009.83. Epub 2009 Apr 21. PMID 19384291
- [Background] Riviere I, Sadelain M. Chimeric Antigen Receptors: A Cell and Gene Therapy Perspective. Mol Ther. 2017 May 3;25(5):1117-1124. doi: 10.1016/j.ymthe.2017.03.034. Epub 2017 Apr 26. PMID 28456379
- [Background] Norelli M, Casucci M, Bonini C, Bondanza A. Clinical pharmacology of CAR-T cells: Linking cellular pharmacodynamics to pharmacokinetics and antitumor effects. Biochim Biophys Acta. 2016 Jan;1865(1):90-100. doi: 10.1016/j.bbcan.2015.12.001. Epub 2015 Dec 31. PMID 26748354
- [Background] Lamers CH, Sleijfer S, van Steenbergen S, van Elzakker P, van Krimpen B, Groot C, Vulto A, den Bakker M, Oosterwijk E, Debets R, Gratama JW. Treatment of metastatic renal cell carcinoma with CAIX CAR-engineered T cells: clinical evaluation and management of on-target toxicity. Mol Ther. 2013 Apr;21(4):904-12. doi: 10.1038/mt.2013.17. Epub 2013 Feb 19. PMID 23423337
- [Background] Till BG, Jensen MC, Wang J, Chen EY, Wood BL, Greisman HA, Qian X, James SE, Raubitschek A, Forman SJ, Gopal AK, Pagel JM, Lindgren CG, Greenberg PD, Riddell SR, Press OW. Adoptive immunotherapy for indolent non-Hodgkin lymphoma and mantle cell lymphoma using genetically modified autologous CD20-specific T cells. Blood. 2008 Sep 15;112(6):2261-71. doi: 10.1182/blood-2007-12-128843. Epub 2008 May 28. PMID 18509084
- [Background] Porter DL, Levine BL, Kalos M, Bagg A, June CH. Chimeric antigen receptor-modified T cells in chronic lymphoid leukemia. N Engl J Med. 2011 Aug 25;365(8):725-33. doi: 10.1056/NEJMoa1103849. Epub 2011 Aug 10. PMID 21830940
- [Background] Turtle CJ, Hanafi LA, Berger C, Gooley TA, Cherian S, Hudecek M, Sommermeyer D, Melville K, Pender B, Budiarto TM, Robinson E, Steevens NN, Chaney C, Soma L, Chen X, Yeung C, Wood B, Li D, Cao J, Heimfeld S, Jensen MC, Riddell SR, Maloney DG. CD19 CAR-T cells of defined CD4+:CD8+ composition in adult B cell ALL patients. J Clin Invest. 2016 Jun 1;126(6):2123-38. doi: 10.1172/JCI85309. Epub 2016 Apr 25. PMID 27111235
- [Background] Davila ML, Riviere I, Wang X, Bartido S, Park J, Curran K, Chung SS, Stefanski J, Borquez-Ojeda O, Olszewska M, Qu J, Wasielewska T, He Q, Fink M, Shinglot H, Youssif M, Satter M, Wang Y, Hosey J, Quintanilla H, Halton E, Bernal Y, Bouhassira DC, Arcila ME, Gonen M, Roboz GJ, Maslak P, Douer D, Frattini MG, Giralt S, Sadelain M, Brentjens R. Efficacy and toxicity management of 19-28z CAR T cell therapy in B cell acute lymphoblastic leukemia. Sci Transl Med. 2014 Feb 19;6(224):224ra25. doi: 10.1126/scitranslmed.3008226. PMID 24553386
- [Background] Mueller KT, Waldron E, Grupp SA, Levine JE, Laetsch TW, Pulsipher MA, Boyer MW, August KJ, Hamilton J, Awasthi R, Stein AM, Sickert D, Chakraborty A, Levine BL, June CH, Tomassian L, Shah SS, Leung M, Taran T, Wood PA, Maude SL. Clinical Pharmacology of Tisagenlecleucel in B-cell Acute Lymphoblastic Leukemia. Clin Cancer Res. 2018 Dec 15;24(24):6175-6184. doi: 10.1158/1078-0432.CCR-18-0758. Epub 2018 Sep 6. PMID 30190371
- [Background] Schuster SJ, Bishop MR, Tam CS, Waller EK, Borchmann P, McGuirk JP, Jager U, Jaglowski S, Andreadis C, Westin JR, Fleury I, Bachanova V, Foley SR, Ho PJ, Mielke S, Magenau JM, Holte H, Pantano S, Pacaud LB, Awasthi R, Chu J, Anak O, Salles G, Maziarz RT; JULIET Investigators. Tisagenlecleucel in Adult Relapsed or Refractory Diffuse Large B-Cell Lymphoma. N Engl J Med. 2019 Jan 3;380(1):45-56. doi: 10.1056/NEJMoa1804980. Epub 2018 Dec 1. PMID 30501490
- [Background] Singh H, Figliola MJ, Dawson MJ, Olivares S, Zhang L, Yang G, Maiti S, Manuri P, Senyukov V, Jena B, Kebriaei P, Champlin RE, Huls H, Cooper LJ. Manufacture of clinical-grade CD19-specific T cells stably expressing chimeric antigen receptor using Sleeping Beauty system and artificial antigen presenting cells. PLoS One. 2013 May 31;8(5):e64138. doi: 10.1371/journal.pone.0064138. Print 2013. PMID 23741305
- [Background] Simon R, Freidlin B, Rubinstein L, Arbuck SG, Collins J, Christian MC. Accelerated titration designs for phase I clinical trials in oncology. J Natl Cancer Inst. 1997 Aug 6;89(15):1138-47. doi: 10.1093/jnci/89.15.1138. PMID 9262252
- [Background] Kershaw MH, Westwood JA, Parker LL, Wang G, Eshhar Z, Mavroukakis SA, White DE, Wunderlich JR, Canevari S, Rogers-Freezer L, Chen CC, Yang JC, Rosenberg SA, Hwu P. A phase I study on adoptive immunotherapy using gene-modified T cells for ovarian cancer. Clin Cancer Res. 2006 Oct 15;12(20 Pt 1):6106-15. doi: 10.1158/1078-0432.CCR-06-1183. PMID 17062687
- [Background] Park JR, Digiusto DL, Slovak M, Wright C, Naranjo A, Wagner J, Meechoovet HB, Bautista C, Chang WC, Ostberg JR, Jensen MC. Adoptive transfer of chimeric antigen receptor re-directed cytolytic T lymphocyte clones in patients with neuroblastoma. Mol Ther. 2007 Apr;15(4):825-33. doi: 10.1038/sj.mt.6300104. Epub 2007 Feb 13. PMID 17299405
- [Background] Kochenderfer JN, Dudley ME, Kassim SH, Somerville RP, Carpenter RO, Stetler-Stevenson M, Yang JC, Phan GQ, Hughes MS, Sherry RM, Raffeld M, Feldman S, Lu L, Li YF, Ngo LT, Goy A, Feldman T, Spaner DE, Wang ML, Chen CC, Kranick SM, Nath A, Nathan DA, Morton KE, Toomey MA, Rosenberg SA. Chemotherapy-refractory diffuse large B-cell lymphoma and indolent B-cell malignancies can be effectively treated with autologous T cells expressing an anti-CD19 chimeric antigen receptor. J Clin Oncol. 2015 Feb 20;33(6):540-9. doi: 10.1200/JCO.2014.56.2025. Epub 2014 Aug 25. PMID 25154820
- [Background] Kochenderfer JN, Dudley ME, Feldman SA, Wilson WH, Spaner DE, Maric I, Stetler-Stevenson M, Phan GQ, Hughes MS, Sherry RM, Yang JC, Kammula US, Devillier L, Carpenter R, Nathan DA, Morgan RA, Laurencot C, Rosenberg SA. B-cell depletion and remissions of malignancy along with cytokine-associated toxicity in a clinical trial of anti-CD19 chimeric-antigen-receptor-transduced T cells. Blood. 2012 Mar 22;119(12):2709-20. doi: 10.1182/blood-2011-10-384388. Epub 2011 Dec 8. PMID 22160384
- [Background] Hay KA, Hanafi LA, Li D, Gust J, Liles WC, Wurfel MM, Lopez JA, Chen J, Chung D, Harju-Baker S, Cherian S, Chen X, Riddell SR, Maloney DG, Turtle CJ. Kinetics and biomarkers of severe cytokine release syndrome after CD19 chimeric antigen receptor-modified T-cell therapy. Blood. 2017 Nov 23;130(21):2295-2306. doi: 10.1182/blood-2017-06-793141. Epub 2017 Sep 18. PMID 28924019
- [Background] Comerota AJ, Throm RC, Miller KA, Henry T, Chronos N, Laird J, Sequeira R, Kent CK, Bacchetta M, Goldman C, Salenius JP, Schmieder FA, Pilsudski R. Naked plasmid DNA encoding fibroblast growth factor type 1 for the treatment of end-stage unreconstructible lower extremity ischemia: preliminary results of a phase I trial. J Vasc Surg. 2002 May;35(5):930-6. doi: 10.1067/mva.2002.123677. PMID 12021709
- [Background] Powell RJ, Simons M, Mendelsohn FO, Daniel G, Henry TD, Koga M, Morishita R, Annex BH. Results of a double-blind, placebo-controlled study to assess the safety of intramuscular injection of hepatocyte growth factor plasmid to improve limb perfusion in patients with critical limb ischemia. Circulation. 2008 Jul 1;118(1):58-65. doi: 10.1161/CIRCULATIONAHA.107.727347. Epub 2008 Jun 16. PMID 18559703
- [Background] Gonin P, Gaillard C. Gene transfer vector biodistribution: pivotal safety studies in clinical gene therapy development. Gene Ther. 2004 Oct;11 Suppl 1:S98-S108. doi: 10.1038/sj.gt.3302378. PMID 15454964
- [Background] Dotti G. T lymphocytes are not immune. Mol Ther. 2013 Jun;21(6):1114-5. doi: 10.1038/mt.2013.102. No abstract available. PMID 23728254
- [Background] Saha S, Woodard LE, Charron EM, Welch RC, Rooney CM, Wilson MH. Evaluating the potential for undesired genomic effects of the piggyBac transposon system in human cells. Nucleic Acids Res. 2015 Feb 18;43(3):1770-82. doi: 10.1093/nar/gkv017. Epub 2015 Jan 20. PMID 25605795
- [Background] Heinrich T, Rengstl B, Muik A, Petkova M, Schmid F, Wistinghausen R, Warner K, Crispatzu G, Hansmann ML, Herling M, von Laer D, Newrzela S. Mature T-cell lymphomagenesis induced by retroviral insertional activation of Janus kinase 1. Mol Ther. 2013 Jun;21(6):1160-8. doi: 10.1038/mt.2013.67. Epub 2013 Apr 23. PMID 23609016
- [Background] Hacein-Bey-Abina S, von Kalle C, Schmidt M, Le Deist F, Wulffraat N, McIntyre E, Radford I, Villeval JL, Fraser CC, Cavazzana-Calvo M, Fischer A. A serious adverse event after successful gene therapy for X-linked severe combined immunodeficiency. N Engl J Med. 2003 Jan 16;348(3):255-6. doi: 10.1056/NEJM200301163480314. No abstract available. PMID 12529469
- [Background] Wang W, Lin C, Lu D, Ning Z, Cox T, Melvin D, Wang X, Bradley A, Liu P. Chromosomal transposition of PiggyBac in mouse embryonic stem cells. Proc Natl Acad Sci U S A. 2008 Jul 8;105(27):9290-5. doi: 10.1073/pnas.0801017105. Epub 2008 Jun 25. PMID 18579772
- [Background] Rad R, Rad L, Wang W, Cadinanos J, Vassiliou G, Rice S, Campos LS, Yusa K, Banerjee R, Li MA, de la Rosa J, Strong A, Lu D, Ellis P, Conte N, Yang FT, Liu P, Bradley A. PiggyBac transposon mutagenesis: a tool for cancer gene discovery in mice. Science. 2010 Nov 19;330(6007):1104-7. doi: 10.1126/science.1193004. Epub 2010 Oct 14. PMID 20947725
- [Background] Fedoroff NV. Presidential address. Transposable elements, epigenetics, and genome evolution. Science. 2012 Nov 9;338(6108):758-67. doi: 10.1126/science.338.6108.758. No abstract available. PMID 23145453
- [Background] Hackett PB, Largaespada DA, Switzer KC, Cooper LJ. Evaluating risks of insertional mutagenesis by DNA transposons in gene therapy. Transl Res. 2013 Apr;161(4):265-83. doi: 10.1016/j.trsl.2012.12.005. Epub 2013 Jan 10. PMID 23313630
- [Background] Zhao S, Jiang E, Chen S, Gu Y, Shangguan AJ, Lv T, Luo L, Yu Z. PiggyBac transposon vectors: the tools of the human gene encoding. Transl Lung Cancer Res. 2016 Feb;5(1):120-5. doi: 10.3978/j.issn.2218-6751.2016.01.05. PMID 26958506
- [Background] Fraietta JA, Lacey SF, Orlando EJ, Pruteanu-Malinici I, Gohil M, Lundh S, Boesteanu AC, Wang Y, O'Connor RS, Hwang WT, Pequignot E, Ambrose DE, Zhang C, Wilcox N, Bedoya F, Dorfmeier C, Chen F, Tian L, Parakandi H, Gupta M, Young RM, Johnson FB, Kulikovskaya I, Liu L, Xu J, Kassim SH, Davis MM, Levine BL, Frey NV, Siegel DL, Huang AC, Wherry EJ, Bitter H, Brogdon JL, Porter DL, June CH, Melenhorst JJ. Determinants of response and resistance to CD19 chimeric antigen receptor (CAR) T cell therapy of chronic lymphocytic leukemia. Nat Med. 2018 May;24(5):563-571. doi: 10.1038/s41591-018-0010-1. Epub 2018 Apr 30. PMID 29713085
- [Background] Milone MC, Bhoj VG. The Pharmacology of T Cell Therapies. Mol Ther Methods Clin Dev. 2018 Jan 31;8:210-221. doi: 10.1016/j.omtm.2018.01.010. eCollection 2018 Mar 16. PMID 29552577
- [Background] Maude SL, Laetsch TW, Buechner J, Rives S, Boyer M, Bittencourt H, Bader P, Verneris MR, Stefanski HE, Myers GD, Qayed M, De Moerloose B, Hiramatsu H, Schlis K, Davis KL, Martin PL, Nemecek ER, Yanik GA, Peters C, Baruchel A, Boissel N, Mechinaud F, Balduzzi A, Krueger J, June CH, Levine BL, Wood P, Taran T, Leung M, Mueller KT, Zhang Y, Sen K, Lebwohl D, Pulsipher MA, Grupp SA. Tisagenlecleucel in Children and Young Adults with B-Cell Lymphoblastic Leukemia. N Engl J Med. 2018 Feb 1;378(5):439-448. doi: 10.1056/NEJMoa1709866. PMID 29385370
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986